CLINICAL TRIAL: NCT04508933
Title: Comparison of Extra Vascular Lung Water Index in Covid-19 ARDS and "Typical"ARDS Patients
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funding
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olcay Dilken, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 0308202247
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Distress Syndrome, Adult; Ventilation Perfusion Mismatch; Pulmonary Edema; Covid19
Keywords: ards; covid19
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Edema; COVID-19; Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Typical ARDS: ARDS due to non Covid19 causes
  Interventions: Device: Extravascular Lung Water Index; Device: Pulmonary Vascular Permeability Index
- C-ARDS: ARDS due to Covid19
  Interventions: Device: Extravascular Lung Water Index; Device: Pulmonary Vascular Permeability Index

INTERVENTIONS:
Device: Extravascular Lung Water Index — Measurement of the EVLWI
Device: Pulmonary Vascular Permeability Index — Measurement of the PVPI

SUMMARY:
Covid-19 also primarily affects endothelium that line up the alveoli. The resulting hypoxemia may differ from "typical" Acute Respiratory Distress Syndrome (ARDS) due to maldistribution of perfusion related to the ventilation. Thus, pathophysiology of Covid-19 ARDS is different, which requires different interventions than typical ARDS. The investigators will assess whether extravascular lung water index and permeability of the alveolar capillary differs from typical ARDS with transpulmonary thermodilution (TPTD) technique. Extravascular Lung Water Index (EVLWI) and Pulmonary Vascular Permeability Index (PVPI) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ARDS defined by Berlin Criteria longer than 24 hours
* Undergoing mechanical ventilation
* Noradrenaline demand >0.1 mcg/kg/min

Exclusion Criteria:

* Not meeting ARDS criteria
* Noninvasive mechanical ventilation
* ARDS resolved shorter than 24 hours
* Shock resolved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ARDS in the adult ICU that have a TPTD catheter inserted since 2018 will be eligible for recruitment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Extravascular Lung Water Index | 1 day
  The amount of fluid accumulated in the lung measured by transpulmonary thermodilution (ml/kg)
Pulmonary vascular permeability index | 1 day
  Integrity of the alveolocapillary barrier measured by transpulmonary thermodilution

CONTACTS AND LOCATIONS:
Overall Officials: Yalım Dikmen, Prof, Study Director — Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data available on reasonable request

REFERENCES:
- [Result] Monnet X, Teboul JL. Transpulmonary thermodilution: advantages and limits. Crit Care. 2017 Jun 19;21(1):147. doi: 10.1186/s13054-017-1739-5. PMID 28625165